CLINICAL TRIAL: NCT06069752
Title: Positional Stability and Refractive Behaviour After In-the-bag Implantation of an Aspheric Hydrophobic IOL After Conventional Phacoemulsification and Femtosecond Laser-Assisted Cataract Surgery
Brief Title: Positional Stability and Refractive Behaviour After Implantation of an IOL After Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Carl Zeiss (Unknown)
Responsible Party: Principal Investigator, Matthias Bolz, Univ.-Prof. Dr., Johannes Kepler University of Linz
Other Study IDs: KUK-Ophthalmology-003
Record Dates: First submitted 2022-08-08; First posted 2023-10-06 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ophthalmological Disorder
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The newest generation Lucia 621 has a step vault design that is claimed to provide excellent positional and refractive predictability.

In order to explore the positional stability, anterior chamber depth stability is examined as marker for haptic buckling comparing positional behaviour after conventional and femtosecond-laser assisted cataract surgery.

DETAILED DESCRIPTION:
In order to explore the positional stability, anterior chamber depth stability is examined as marker for haptic buckling comparing positional behaviour after conventional and femtosecond-laser assisted cataract surgery.

Furthermore, the refractive outcome of CT Lucia 621P/PY is examined, providing optimized (en bloc optimization) formula constants for both, conventional and femtosecond-laser assisted cataract surgery for Haigis, Hoffer Q, Holladay I, SRK/T and Castrop formulae.

Besides ACD, further parameters for IOL stability are examined (IOL tilt/decentration) and consequences for the aberration profile are described.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject with a minimum age of 22 years
* Planned natural lens replacement with posterior chamber IOL implantation
* Clear intraocular media other than cataract
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visit
* Ability to consent to the participation in study
* Signed informed consent

Exclusion Criteria:

* Corneal pathology/ectasia
* Prior ophthalmic surgery
* Zonular-defects, unstable bag
* Macular pathologies
* Expected Visual acuity of less than 0.63 (decimal)
* Glaucoma
* Use of systemic or ocular medication that might affect vision
* Patient is pregnant, plans to become pregnant, is lactating
* Concurrent participation in any other clinical trial with an investigation product

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 50 subjects requiring IOL implantation to treat aphakia after extracapsular cataract extraction or phacoemulsification.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Tilt and decentration of intraocular lens measured in degrees | 1 month post surgery compared with 12 months post surgery
  Tilt and decentration of intraocular lens measured in degrees with Casia-2 Anterior Segment Optical Coherence Tomography 1 month post surgery compared with 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Principal Investigator — JKU Linz
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casazza M, Reifeltshammer SA, Hirnschall N, Mariacher S, Laubichler P, Siska R, Wendelstein J, Bolz M. Randomized controlled bilateral comparison of femtosecond laser-assisted cataract surgery versus conventional phacoemulsification. BMJ Surg Interv Health Technol. 2025 Jul 10;7(1):e000342. doi: 10.1136/bmjsit-2024-000342. eCollection 2025. PMID 40662090